CLINICAL TRIAL: NCT06425939
Title: Exploring the Relationship Between Heart Rate Variability (HRV), Training Load, and Exercise Performance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PEP-2401
Record Dates: First submitted 2024-05-16; First posted 2024-05-23 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Heart Rate Variability; Exercise
Keywords: exercise performance; HRV; training load; Whoop; wrist worn tracker; exercise recovery
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (Other): Healthy adults moderately trained in resistance exercises
  Interventions: Other: Force plate assessment; Device: Whoop wrist band

INTERVENTIONS:
Other: Force plate assessment — On Day 1, Day 45 and Day 90: 3x drop jumps, 2 min rest, 3x counter movement jumps, 2 min rest, 3x dynamic push-ups
Device: Whoop wrist band — Whoop wrist worn activity tracker (not a medical device) collects continuous data via smartphone app. This is a marketed device. This is not a device study.

SUMMARY:
Heart rate variability (HRV) is a measure of the variation in time between each heartbeat.

It is an indirect and ubiquitous biomarker of performance readiness and recovery measured by most consumer-grade wearable fitness trackers. However, there is little documented on the relationship between HRV, training load, and performance measures in the Real-World.

Whoop wrist-worn activity trackers have been validated against the gold-standard Electrocardiography (ECG) for HRV and HR measurements. Whoop leverages photoplethysmography (PPG) technology to continuously track (HR, HRV, respiratory rate, energy expenditure) and provides, daily, individual insights, trends, and coaching to improve strain, sleep, and recovery. Research has demonstrated that heart rate variability (HRV) guided training may be more optimal compared to predetermined training for aerobic exercise improvements.

The purpose of this study is to assess the feasibility of providing personalized training recommendations based on HRV measured by a consumer-grade wearable (Whoop) in a real-world setting to better understand the HRV relationship with performance.

DETAILED DESCRIPTION:
The purpose of this study is to determine if Training Intensity (%HRmax in min.) during Low HRV periods acutely (below HRV baseline next day and consecutive days) and chronically (weeks below previous weeks HRV baseline) will have a negative relationship with Post-Test Performance Metrics as measured by Force Plates, which could lead to personalized training recommendations using HRV. The Investigators conducted a pilot study using Whoop devices to monitor 50 subjects for 3 months and observed that individuals had High Training Load (above their baseline) on Low HRV days (below their baseline) on over 200 days. The Investigators hypothesize seeing similar High Training Load on Low HRV days during this study and would like to understand that relationship with Performance

Primary objective: To determine if Training Intensity (%HRmax in min.) during Low HRV periods acutely (below HRV baseline next day and consecutive days) and chronically (weeks below previous weeks HRV baseline) will have a negative relationship with Post-Test Performance Metrics as measured by Force Plates.

Secondary Objective : Measure and determine if subjective journal entries (mood, anxiety, recovery, etc.) are related to HRV, RHR, Sleep Quantity, and Sleep Efficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Actively participating in resistance training 2-4 times per week.
2. Age 21-50 years, male and female.
3. Subject is willing to refrain from vigorous exercise (light physical activity only) 24 hours prior to visit(s).
4. Subject is willing to avoid alcohol consumption 24 hours prior to visit(s).
5. Subject is willing to provide consent.
6. Subject is able to continuously wear a wrist-worn device, including during sleep, except when submerged underwater (i.e., swimming, bathing).

Exclusion Criteria:

1. Individual has a condition the Investigator believes would interfere with his ability to provide informed consent, comply with the project/study protocol, which might confound the interpretation of the project/study results or put the person at undue risk.
2. Those with a medical history that would interfere with the results of this study.
3. Under the care of a physician.
4. Skin sensitivities.
5. Sleep disorders.
6. Using prescription medications that would impact sleep.
7. If female, you are not pregnant, planning to get pregnant or currently breast feeding.
8. Smoker.
9. Not able to wear wrist-worn device continuously.
10. Lack of proficiency in English.
11. Lack of proficiency or access to the internet and email address.
12. Participation in another clinical trial within the past 30 days.
13. Subject is employed by, or has a parent, guardian, or other immediate family member employed by a company that manufactures any products that compete with any Gatorade product. If subject is unsure if a company would be considered a competitor to Gatorade, they will be asked to please let the study investigator know the name of the other company and the nature of their relationship to that company before they sign the informed consent.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Training Intensity | Change from baseline (Day 1) to mid-study (Day 45) and end of study (Day 90)
  % HRmax (in minutes) measured by force plates
Performance | Change from baseline (Day 1) to mid-study (Day 45) and end of study (Day 90)
  Reactive Strength Index in cm/s using force plates
Peak Power Output | Change from baseline (Day 1) to mid-study (Day 45) and end of study (Day 90)
  W/kg using force plates
Jump Height | Change from baseline (Day1) to mid-study (Day 45) and end of study (Day 90)
  (cm) using force plates
Dynamic Push Ups Peak Force | Change from baseline (Day 1) to mid-study (Day 45) and end of study (Day 90)
  (N)) using force plates

SECONDARY OUTCOMES:
Correlation of subjective measures to Heart Rate Variability (HRV) | Daily for 90 days
  True or False answers to Whoop app journal questions for mood, e.g., nervous, anxious, stability, motivation, energy, feeling sick or stressed, hydration, recovery, consumption of alcohol, caffeine, or melatonin
Correlation of subjective measures to resting heart rate (RHR) | Daily for 90 days
  True or False answers to Whoop app journal questions for mood, e.g., nervous, anxious, stability, motivation, energy, feeling sick or stressed, hydration, recovery, consumption of alcohol, caffeine, or melatonin
Correlation of subjective measures to sleep quantity | Daily for 90 days
  True or False answers to Whoop app journal questions for mood, e.g., nervous, anxious, stability, motivation, energy, feeling sick or stressed, hydration, recovery, consumption of alcohol, caffeine, or melatonin
Correlation of subjective measures to sleep efficiency | Daily for 90 days
  True or False answers to Whoop app journal questions for mood, e.g., nervous, anxious, stability, motivation, energy, feeling sick or stressed, hydration, recovery, consumption of alcohol, caffeine, or melatonin

CONTACTS AND LOCATIONS:
Overall Officials: Corey Ungaro, PhD, Principal Investigator — PepsiCo, Inc. Sports Science
Locations (2):
- United States (2):
  - PepsiCo R&D, Gatorade Sports Science Institute, Chicago, Illinois
  - PepsiCo R&D, Gatorade Sports Science Institute, Frisco, Texas

IPD SHARING:
Plan to Share IPD: No